CLINICAL TRIAL: NCT04069455
Title: A Randomized, Multi-center, Prospective Study Evaluating e-Patient Report Outcomes (ePRO) for Adjuvant Chemotherapy in Chinese Patients With Colorectal Cancers
Brief Title: ePRO for Adjuvant Therapy of Colorectal Adenocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Principal Investigator, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRCCZ-ePRO2
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Carcinoma
Keywords: electronic patient reported outcomes; colorectal carcinoma; adjuvant chemotherapy; quality of life
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPRO group (Experimental): Clinical usual care plus ePRO App self-management online during postoperative adjuvant chemotherapy
  Interventions: Other: Electronic Patients Reported Outcomes
- Control group (No Intervention): Clinical usual care during postoperative adjuvant chemotherapy

INTERVENTIONS:
Other: Electronic Patients Reported Outcomes — ePRO is a application which is web based and accessible from home or mobile device, for patients to complete symptom reports and receive severity-based advice
  Other Names: ePRO
  Arms: EPRO group

SUMMARY:
It is a multi-centric randomized controlled trial. The goal of this study is to observe the improvement of QoL using ePRO to manage patients with colorectal cancer who received Oxaliplatin-based adjuvant chemotherapy.The prognosis will also be studied.

DETAILED DESCRIPTION:
The most of advanced colorectal carcinoma are underwent postoperative chemotherapy. Adverse events (AE) during chemotherapy disrupt treatment and impair the patients' quality of life(QoL). Under usual care, the patients are largely required to self-monitor symptoms at home. Patients can lack confidence in making decisions between obtaining clinical support or self-managing and can delay seeking medical advice, heightening the risk of symptom escalation and hospital admissions and impact the efficacy of chemotherapy finally. There is growing evidence that the utilisation of patient-reported outcome(PRO) measures can aid the timely identification of physical and psychosocial disorders, facilitate patient-doctor communication and assist decision-making. There has been a drive to develop electronic systems(ePRO) to allow remote real-time patient monitoring during cancer therapy. Positive patient benefit (including QOL and survival) was recently reported in a US trial of an online system for metastatic cancer treatment.

The trial is a prospective randomised two-arm parallel group design study with repeated measures and mixed methods. Participants (adult patients with colorectal cancer on adjuvant chemotherapy) are randomised to receive the ePRO intervention or usual care over 24 weeks of treatment. Participants in the intervention arm receive training in using the ePRO APP system to provide routine weekly adverse event reports from home. Hospital staff can access ePRO reports via APP and use the information during consultations or phone calls or message with patients. The overall target sample for the trial is N = 270. The primary outcome of is quality of life (EORTC QLQ-C30/CR29) with secondary outcomes including the proportion of completed chemotherapy, AE, DFS, OS and patient self-efficacy. Outcome data is collected at baseline, 3, 6 and 12 months. The intervention is also being evaluated via end of study interviews with patient participants and clinical staff.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old (inclusive), regardless of gender.
2. Patients with colorectal cancer diagnosed by cytology or histopathology.
3. The patient underwent radical surgery for cancer. Radical surgery is defined as routine laparotomy or laparoscopic radical surgery for the purpose of radical
4. The ECOG performance status is 0 to 2 points and able to receive adjuvant chemotherapy.
5. Patients must be randomized within 2 months after the surgery.
6. According to the investigator's judgment, the patient has recovered from surgical side effects after radical surgery (e.g., the wound has healed fully without complications).
7. Oxaliplatin regimen is planned to be used for postoperative adjuvant chemotherapy for 3 to 6 months
8. The blood pregnancy test results of women of childbearing age must be negative within 7 days prior to randomization.
9. The main organs function well. That is, the relevant inspection indexes within 14 days prior to enrollment meet the following requirements:

   a) Routine blood test: i. Leukocyte≥ 4.0×109/L; ii. Neutrophil count > 1.5×109/L; iii. Blood platelet count > 80×109/L; iv. Hemoglobin > 90 g/L (No blood transfusion in 14 days); b) Biochemistry test: i. TBil ≤ 1.5×ULN (upper limit of normal); ii. Blood glutamic alanine aminotransferas (ALT) or serum aspartate aminotransferase (AST) ≤ 2.5×ULN; iii. Endogenous creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula); c) Cardiac doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ 50%.
10. The patient has provided written informed consent prior to any study-specific procedures, and is willing and able to be present during the study and follow the study procedure during treatment and follow-up.

Exclusion Criteria:

1. <18 years old or >75 years old.
2. Other tumors except gastric and colorectal cancer.
3. Metastasis has occurred.
4. Female during pregnancy or lactation.
5. A history of other malignant tumors within 5 years, except for adequately treated basal cell carcinoma or squamous cell carcinoma or carcinoma in situ.
6. The patient is known to be allergic to oxaliplatin, 5-FU, folinic acid or any excipients of these products.
7. Evidence of any severe or uncontrolled systemic disease, including but not limited to:

   1. Unstable or decompensated respiratory, cardiac, liver or kidney disease;
   2. HIV infection;
   3. Uncontrol high blood pressure, diabetes;
   4. Severe arrhythmia;
   5. Massive active bleeding.
8. A history of alcohol abuse or drug abuse.
9. As judged by the investigator, there is a low likelihood of enrollment (including inability to understand study requirements, poor compliance, infirmity, inability to ensure that the protocol can be followed as required, etc.), or there are other factors considered by the investigator to be unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Global health and functional scores | 6 months after surgery
  Global health and functional scores will be evaluated by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 version 3.0 (EORTC QLQ-C30) questionnaire.It comprises a two-item global health status domain and five multi-item functional domains (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning); Items were scaled and scored according to the EORTC Scoring Manual. Raw scores were transformed to a linear scale ranging from 0 to 100. For scores measuring global health status and functional domains, a higher score represents a 'better' level of status or functioning.
C30 symptom scores | 6 months after surgery
  C30 symptom scores will be evaluated by EORTC QLQ-C30 questionnaire. It comprises three multi-item symptom domains (fatigue, pain, and nausea and vomiting); and six single-item domains for the assessment of additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and the perceived financial impact of the disease and treatment. Items were scaled and scored according to the EORTC Scoring Manual. Raw scores were transformed to a linear scale ranging from 0 to 100. A higher score for symptom domains represents a 'worse' level of symptoms.
CR29 scores | 6 months after surgery
  CR29 scores will be evaluated by European Organization for Research and Treatment of Cancer (EORTC) questionnaire module for colorectal cancer, the QLQ-CR29. It was created with six hypothesised scales (micturition, pain, faecal incontinence, defaecation problems, anxiety and body image) and 11 single items. Raw scores were transformed to a linear scale ranging from 0 to 100.a high score for a symptom scale represents a high level of symptomatology or problems.

SECONDARY OUTCOMES:
the incidence of adverse events | baseline, 3, 6 and 12 months after surgery
  AE
the proportion of completed chemotherapy | 3 and 6 months after surgery
Disease free survival | 36 months after randomized
  DFS
Overall survival | 36 months after randomized
  OS

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, MD, Principal Investigator — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- GuoXiang Cai, Shanghai, Shanghai Municipality, China